CLINICAL TRIAL: NCT02121782
Title: A Randomized, Open-label (Part A) or Double-blind (Part B), Active-controlled (Part B) Phase I/IIa Study to Investigate the Safety, Tolerability, and Immunogenicity of GC3110A (Quadrivalent Influenza Vaccine)
Brief Title: A Phase I/IIa Study of GC3110A (Quadrivalent Influenza Vaccine)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC3110A_P1/2a
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Influenza
Keywords: QIV; Quadrivalent Influenza Vaccine; Influenza vaccine; Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Quadrivalent influenza vaccine(Part A) (Experimental): Day 1: GC3110A, 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Quadrivalent influenza vaccine
- Quadrivalent influenza vaccine(Part B) (Experimental): Day 1: GC3110A, 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Quadrivalent influenza vaccine
- Trivalent influenza vaccine(Part B) (Active Comparator): Day 1: GC Flu Pre-filled Syringe Inj., 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Trivalent influenza vaccine

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — GC3110A, 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC3110A
  Arms: Quadrivalent influenza vaccine(Part A); Quadrivalent influenza vaccine(Part B)
Biological: Trivalent influenza vaccine — GC Flu Pre-filled Syringe Inj., 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC Flu Pre-filled Syringe Inj.
  Arms: Trivalent influenza vaccine(Part B)

SUMMARY:
The purpose of this study is to determine whether GC3110A (a QIV) is effective compared to GC Flu Pre-filled Syringe Inj. (a marketed TIV) after single intramuscular administration in Korean healthy adults.

The comparator, GC Flu pre-filled syringe inj. is a trivalent influenza vaccine (TIV) including viruses representing 3 influenza strains (one A/HIN1, one A/H3N2, and one B). However, two antigenically distinct lineages of influenza B (Victoria and Yamagata) co-circulate annually in the United States. Predicting which lineage of influenza B will predominate during a season is challenging, and cross-protection by immunization against the other lineage is expected to be low. One proposed alternative is to produce a quadrivalent influenza vaccine (QIV) including an influenza B virus from each of the two circulating lineages. GC3110A is a new quadrivalent influenza vaccine (QIV), which contains all of 4 vaccine components WHO recommends for use in the 2013-14 influenza season (northern hemisphere winter) and includes two influenza B viruses. GC3110A is expected to show the additional public health benefit compared with traditional TIV.

DETAILED DESCRIPTION:
This study is the first in human trial of GC3110A and is designed as an adaptive Phase I/IIa to ensure participants protection. Part A is an open-label and single arm study in 9 healthy volunteers. Data and Safety Monitoring Board (DSMB) will review the solicited/unsolicited adverse events conditionally if any toxicity of Grade 3 or 4 has been reported during 7 days after vaccination. Part B is a randomized (2:1), double-blind, active controlled study and a total of 75 volunteers will participate in this part. Adverse events assessment will be done according to the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials'.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Healthy Korean adults (age: between over 19 and under 65)
* Korean adults who agree with 21 days follow up after vaccination and good compliance to study procedures
* Those who are able to comply with the requirements for the study

Exclusion Criteria:

* Inability in written/verbal communication
* Subjects who have participated in other interventional study within 30 days
* Alcohol or drug abuse within 6 months
* Heavy drinkers or subjects who do not agree to stop drinking for 3 days before vaccination and other 3 days after vaccination
* Who got the treatment of psychotropic drugs and narcotic analgesic drugs within 6 months of enrollment
* Hypersensitivity with drug or active ingredient
* Disorders in immune function
* History of Guillain-Barré syndrome
* Disease/medications which are likely to cause any severe bleeding
* Active infection or experience of fever (>38.0 ℃) within 72 hours following vaccination
* Oral temperature >38.0 ℃ at the vaccination day
* Erythema, tattoo, injury at shoulder (vaccination site)
* Hypersensitivity with egg, chicken, or any of the vaccine components, or Neomycin, Gentamicin
* Influenza vaccination within 6months
* Any vaccination within 30 days
* Concomitant medications/therapy such as immunosuppressants or immune modifying drugs, systemic corticosteroids, immunoglobulins, blood or blood- derived products, or anti-cancer chemotherapy or radiation therapy within3 months
* Pregnant or breast-feeding women
* Clinically significant underlying diseases or medical history at investigator's discretion

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events following vaccination | Day 1 up to 7 Days post vaccination
  Solicited injection site reactions: Pain, Tenderness, Erythema, Redness, Induration, and Swelling; Solicited systemic reactions: Fever, Sweating, Chill, Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, arthralgia.
Unsolicited adverse events following vaccination | Day 1 up to 22 Days post vaccination
  It can be estimated by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials
Seroconversion rate of HI (Hemagglutination Inhibition) antibody for each strain | Day 22 post vaccination
Seroprotection rate of HI (Hemagglutination Inhibition) antibody for each strain | Day 22 post vaccination

SECONDARY OUTCOMES:
Abnormalities in physical examination, vital signs, and/or clinical laboratory tests | Day 22 post vaccination
GMT(geometric mean titers) for each strain | Day 22 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo KIM, M.D., Ph.D., Principal Investigator — Korea University Guro Hospital; Chang-Hee Lee, M.D., Study Director — Green Cross Corporation
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea